CLINICAL TRIAL: NCT04809883
Title: Normative EndoFlip Data on the Diameter and Distensibility of the Pylorus During Fasting and Postprandially in Healthy Females and Male Adults
Brief Title: A Study to Evaluate Endoflip Normal Ranges Data in Healthy Volunteers
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Michael Camilleri, MD, Principal Investigator, Mayo Clinic
Other Study IDs: 20-012285
Record Dates: First submitted 2021-03-02; First posted 2021-03-22 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- observational study of gastric and pyloric motor function measured with Endoflip: observational study of gastric and pyloric motor function measured with Endoflip during fasting and postprandial periods There is NO intervention
  Interventions: Diagnostic Test: Endoflip measurement of gastric and pyloric function

INTERVENTIONS:
Diagnostic Test: Endoflip measurement of gastric and pyloric function — Endoflip device to measure gastric and pyloric functions

SUMMARY:
The purpose of this research is to establish the normal range of diameter and distensibility of pylorus and the fasting and postprandial antro-pyloric motility in healthy adults.

DETAILED DESCRIPTION:
An Endoflip catheter will be placed through the mouth into the stomach in order to measure distal antral contractile activity and pyloric diameter and distensibility during fasting and after the ingestion of a standard meal

ELIGIBILITY:
Inclusion Criteria:

* Females and males.
* Between the ages of 18 and 65 years.
* Body mass index between 18 and 35 kg/m^2.

Exclusion Criteria:

* Heartburn, regurgitation, or symptoms suggestive of gastroparesis such as nausea, early satiety, postprandial bloating, and upper abdominal pain.
* Pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — equal number of males and females will be recruited for this study in up to 45 adults
Study Population: healthy adults between the ages of 18 and 65 with body mass indices between 18 and 35 kilograms/meter squared will be recruited for this study
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-03-06 (Actual); Primary Completion 2021-06-23 (Actual); Study Completion 2021-06-23 (Actual)

PRIMARY OUTCOMES:
fasting and postprandial pyloric diameter | 1 hour prior to meal and 1 hour following standardized meal
  Change in Pyloric diameter will be measured during fasting and postprandial using Endoflip
fasting and postprandial pyloric distensibility index | 1 hour prior to meal and 1 hour following standardized meal
  Change in Pyloric distensibility index will be measured during fasting and postprandial using Endoflip
fasting and postprandial distal antral motility index | 1 hour prior to meal and 1 hour following standardized meal
  Change in distal antral motility index will be measured during fasting and postprandial using Endoflip

CONTACTS AND LOCATIONS:
Overall Officials: Michael Camilleri, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Michael Camilleri, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials